CLINICAL TRIAL: NCT04002934
Title: A Phase II Randomized, Double-Blind, Parallel-Group, Placebo Controlled Delayed-Start Trial to Assess the Efficacy, Safety, and Tolerability of Bazedoxifene Acetate (BZA) as a Remyelinating Agent in Patients With Multiple Sclerosis
Brief Title: Bazedoxifene Acetate as a Remyelinating Agent in Multiple Sclerosis
Acronym: ReWRAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Riley Bove, MD (Other)
Responsible Party: Sponsor-Investigator, Riley Bove, MD, Assistant Professor of Neurology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ReWRAP; 138495 (Other: FDA -- Investigational New Drug Number); 18-24511 (Other: UCSF IRB No.)
Record Dates: First submitted 2019-06-25; First posted 2019-07-01 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting
Keywords: MS; RRMS; Remyelination; Repair; Multiple Sclerosis; SERM; Estrogen; BZA; Bazedoxifene; Myelin Repair; Conbriza
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — bazedoxifene

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo controlled, double-blind, delayed-start trial of BZA in 50 women with MS to be given as follows:
  Group A will receive 3 months of BZA + 3 months of BZA; Group B will receive 3 months of placebo + 3 months of BZA
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A is the "early-start" group and will receive a total of 6 months of BZA -- 3 months of BZA, followed by 3 months BZA
  Interventions: Drug: Bazedoxifene Acetate
- Group B (Experimental): Group B is the "delayed-start" group and will receive a total of 3 months of BZA -- 3 months of placebo, followed by 3 months of BZA
  Interventions: Drug: Bazedoxifene Acetate

INTERVENTIONS:
Drug: Bazedoxifene Acetate — 40 mg Bazedoxifene delivered orally in the form of 2x 20 mg blinded capsules
  Other Names: Bazedoxifene; Conbriza; Viviant; TSE-424; WAY 140424; WAY-140424

SUMMARY:
The primary goal of this study is to assess the efficacy of bazedoxifene (BZA) as remyelinating agent in patients with relapsing-remitting multiple sclerosis (RRMS).

The investigators will utilize electrophysiologic techniques and magnetic resonance imaging to quantify the effect of treatment in 50 women over the course of 6 months.

Participants may remain on their standard disease modifying treatment during the course of the trial but may not concurrently participate in any other investigational new drug research study.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic neurologic disorder characterized by the loss of myelin, which results in disruption of nerve signal, damage to axons, and, ultimately, neurodegeneration. In order to treat MS, new methods for promoting repair (remyelination) are sorely needed.

There is a strong preclinical (including EAE) and epidemiologic rationale for investigating the remyelinating potential of estrogenic compounds, including evidence of endogenous (puberty, postpartum periods) and exogenous hormonal influences on MS risk and course. MS affects 3 times more women than men, and disease course in women appears overall less aggressive (on MRI, fewer T2-hyperintense demyelinated lesions develop into axonal destruction visualized as hypointense T1 "black holes").

Bazedoxifene (BZA), a third-generation SERM with extensive safety data in humans, was identified in a novel high-throughput screen (BIMA screen) for compounds capable of promoting remyelination. Subsequent analysis validated BZA's remyelinating effect in vitro and in vivo following demyelinating insult. Given strong pre-clinical support for BZA's remyelinating potential, and the clinical success of other compounds identified using the BIMA screen (Green et al., 2017), the investigators will investigate the use of BZA as a remyelinating therapy in patients with MS.

ELIGIBILITY:
Expanded Inclusion Criteria:

1. Relapsing remitting Multiple Sclerosis by 2017 Revised McDonald Criteria
2. Women aged 45-65 or 40+ post-menopausal.
3. Stable immunomodulatory therapy - no switch or planned switch in < 6 months and no change in doses in 30 days prior to screening
4. Use of contraceptive method with ≤1% failure rate during period of trial if premenopausal
5. Understand and sign informed consent.
6. EDSS 0-6.0 (inclusive)

Chronic Optic Neuropathy Subgroup Inclusion Criteria (including broader inclusion criteria):

1. Expanded inclusion criteria
2. Latency delay > 118 milliseconds on baseline full-field transient pattern reversal VEP in at least one eye (electrophysiological evidence of demyelination)

Expanded Exclusion Criteria:

1. Multiple Sclerosis disease duration > 25 years
2. History of significant cardiac conduction block
3. Patients with a known, suspected or past history of breast, gynecological, or gastrointestinal cancer
4. Suicidal ideation or behavior in 6 months prior to baseline
5. Pregnancy, breastfeeding, or planning to become pregnant
6. Included with other study protocol simultaneously without prior approval
7. Concomitant or prior use of any other putative remyelinating therapy as determined by investigator, including but not limited to Clemastine, Duavee, and Tamoxifen.
8. Serum creatinine > 1.5mg/dL; AST, ALT, or alkaline phosphatase > 2 times the upper limit of normal
9. History of drug or alcohol abuse within the past year
10. Untreated B12 deficiency (as determined by B12 serological assessments and metabolites including methylmalonic acid [MMA] and homocysteine) or untreated hypothyroidism
11. Clinically significant cardiac, metabolic, hematologic, hepatic, immunologic, urologic, endocrinologic, neurologic, pulmonary, psychiatric, dermatologic, allergic, renal or other major diseases that in the PI's judgement may affect interpretation of study results or patient safety.
12. History of or presence of clinically significant medical illness or laboratory abnormality that, in the opinion of the investigator would preclude participation in the study.
13. Patients whose lack of mobility exposes them to an increased risk of venous thromboembolism
14. Patients with undiagnosed uterine bleeding
15. Patients with unknown, suspected or past history of breast cancer
16. Patients with known or suspected estrogen-dependent neoplasia
17. Patients with active or a past history of venous thromboembolism
18. Patients with active or a past history of arterial thromboembolism
19. Patients with known protein C, protein S, or antithrombin deficiency or other known thrombophilic disorders
20. Patients with hypersensitivity (angioedema, anaphylaxis) to estrogens, bazedoxifene, or any ingredients
21. Patients with known hepatic impairment or disease

Chronic Optic Neuropathy Subgroup Exclusion Criteria:

1. Expanded exclusion criteria
2. Optic neuritis in prior 6 months
3. Known optic neuritis in involved eye ≥ 15 years ago
4. Major ophthalmologic disease/Concomitant ophthalmologic disorders (e.g. diabetes, macular degeneration, glaucoma, severe myopia, etc.).
5. Myopia > -7 Diopters (severe myopia)
6. Disc hemorrhages in qualifying eye
7. No light perception in qualifying eye
8. Simultaneous bilateral optic neuritis
9. Cotton wool spots in qualifying eye
10. Macular star in qualifying eye

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Myelin Water Fraction (MWF) on MRI | 3 months
  The primary objective is to evaluate the efficacy of BZA relative to placebo for increasing MWF on MRI within normal appearing white matter of the corpus callosum, between baseline and 90 days in a double-blinded trial (1st 90 days in the early start group versus 1st 90 days of the delayed start group).

SECONDARY OUTCOMES:
Changes in BICAMS scores | 3 months
  The first key secondary objective is changes in BICAMS scores over 3 months.
Changes in MSFC scores | 3 months
  The second key secondary objective is changes in MSFC scores over 3 months.
Changes in BICAMS scores | 6 months
  The third key secondary objective is changes in BICAMS scores over 6 months.
Changes in MSFC scores | 6 months
  The fourth key secondary objective is changes in MSFC scores over 6 months.
Myelin Water Fraction (MWF) on MRI | 6 months
  The fifth key secondary objective is to assess whether MWF at 180 days increases to a greater extent in the early start group (exposed to BZA for 90 days during both Stage 1 and Stage 2) when compared to the delayed start group (exposed to placebo during Stage 1 and BZA for only 90 days during Stage 2).
Visual Evoked Potential (VEP) P100 Latency | 3 months
  The sixth key secondary objective is changes in visual evoked potential (VEP) P100 latency.
Visual Evoked Potential (VEP) P100 Latency | 6 months
  The seventh key secondary objective is changes in visual evoked potential (VEP) P100 latency.
Novel Digital Measures of Cognition | 6 months
  The eighth key secondary objective is to assess novel digital measures of cognition (processing speed from EVO Monitor).
FitBit Activity | 6 months
  The ninth key secondary objective is to assess daily activity by average daily step count as well as sleep activity by various sleep metrics recorded through FitBit.
Serum Neurofilament Light Chain (NFL) levels | 6 months
  The tenth key secondary objective is to assess NFL levels.
Expanded Disability Status Scale (EDSS) | 6 months
  The last key secondary objective is an assessment of exploratory outcomes, including EDSS.
Bladder Control Scale (BLCS) | 6 months
  The last key secondary objective is an assessment of exploratory outcomes, including the BLCS, a patient-reported outcome.
Bowel Control Scale (BWCS) | 6 months
  The last key secondary objective is an assessment of exploratory outcomes, including the BWCS, a patient-reported outcome.
Pittsburgh Sleep Quality Index (PSQI) | 6 months
  The last key secondary objective is an assessment of exploratory outcomes, including the PSQI, a patient-reported outcome.
12-Item Multiple Sclerosis Walking Scale (MSWS-12) | 6 months
  The last key secondary objective is an assessment of exploratory outcomes, including the MSWS-12, a patient-reported outcome.
Center for Epidemiological Studies Depression Scale (CESD) | 6 months
  The last key secondary objective is an assessment of exploratory outcomes, including the CESD, a patient-reported outcome.
Modified Fatigue Impact Score (MFIS) | 6 months
  The last key secondary objective is an assessment of exploratory outcomes, including the MFIS, a patient-reported outcome.
36-Item Short Form Survey (SF36) | 6 months
  The last key secondary objective is an assessment of exploratory outcomes, including the SF36, a patient-reported outcome. , Visual Function Questionnaire (VFQ25); other MRI metrics, including total volume of T2 lesions, number of new/enlarging T2 lesions, atrophy in corpus callosum, thalamus, prefrontal cortex, and other exploratory structures; Timed Up and Go test; and FitBit measures of variability in step count.
Visual Function Questionnaire (VFQ25) | 6 months
  The last key secondary objective is an assessment of exploratory outcomes, including the VFQ25, a patient-reported outcome.
Total T2 Lesion Volume | 6 months
  The last key secondary objective is an assessment of exploratory outcomes, including total volume of T2 lesions.
Number of New/Enlarging T2 Lesions | 6 months
  The last key secondary objective is an assessment of exploratory outcomes, including the number of new/enlarging T2 lesions.
Levels of Brain Atrophy | 6 months
  The last key secondary objective is an assessment of exploratory outcomes, including levels of atrophy in the corpus callosum, thalamus, prefrontal cortex, and other exploratory structures.
Timed Up and Go (TUG) test | 6 months
  The last key secondary objective is an assessment of exploratory outcomes, including the TUG test.

OTHER OUTCOMES:
Tolerability and Safety of BZA - Patient Hot Flash Diary | 6 months
  The tertiary objectives are to demonstrate the tolerability and document the safety of BZA in this population of patients. Tolerability and safety of BZA will be assessed by patient hot flash diaries.
Tolerability and Safety of BZA - Treatment Satisfaction Questionnaire for Medication (TSQM) | 6 months
  The tertiary objectives are to demonstrate the tolerability and document the safety of BZA in this population of patients. Tolerability and safety of BZA will be assessed by the Treatment Satisfaction Questionnaire for Medication (TSQM).
Tolerability and Safety of BZA - Patient Reports of Spasms | 6 months
  The tertiary objectives are to demonstrate the tolerability and document the safety of BZA in this population of patients. Tolerability and safety of BZA will be assessed by patient reports of spasms.
Tolerability and Safety of BZA - Safety Monitoring Labs | 6 months
  The tertiary objectives are to demonstrate the tolerability and document the safety of BZA in this population of patients. Tolerability and safety of BZA will be assessed by safety monitoring labs.
Tolerability and Safety of BZA - Records of Adverse Events | 6 months
  The tertiary objectives are to demonstrate the tolerability and document the safety of BZA in this population of patients. Tolerability and safety of BZA will be assessed by records of adverse events.
Tolerability and Safety of BZA - Monitoring MS Relapses | 6 months
  The tertiary objectives are to demonstrate the tolerability and document the safety of BZA in this population of patients. Tolerability and safety of BZA will be assessed by monitoring MS relapses throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Riley M Bove, MD MMSc, Principal Investigator — University of California, San Francisco
Locations (1):
- Weill Institute for Neurosciences, University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Green AJ, Gelfand JM, Cree BA, Bevan C, Boscardin WJ, Mei F, Inman J, Arnow S, Devereux M, Abounasr A, Nobuta H, Zhu A, Friessen M, Gerona R, von Budingen HC, Henry RG, Hauser SL, Chan JR. Clemastine fumarate as a remyelinating therapy for multiple sclerosis (ReBUILD): a randomised, controlled, double-blind, crossover trial. Lancet. 2017 Dec 2;390(10111):2481-2489. doi: 10.1016/S0140-6736(17)32346-2. Epub 2017 Oct 10. PMID 29029896
- [Derived] Nylander A, Anderson A, Rowles W, Hsu S, Lazar AA, Mayoral SR, Pease-Raissi SE, Green A, Bove R. Re-WRAP (Remyelination for women at risk of axonal loss and progression): A phase II randomized placebo-controlled delayed-start trial of bazedoxifene for myelin repair in multiple sclerosis. Contemp Clin Trials. 2023 Nov;134:107333. doi: 10.1016/j.cct.2023.107333. Epub 2023 Sep 20. PMID 37739167
- [Derived] Morales-Rodriguez D, Anderson A, Nylander A, Hsu S, Singh J, Rowles W, Walsh CM, Braley TJ, Bove R. Well-being at midlife: Correlates of mental health in ambulatory menopausal women with multiple sclerosis. Mult Scler. 2023 Oct;29(11-12):1493-1502. doi: 10.1177/13524585231197056. Epub 2023 Sep 16. PMID 37715710
- See also: Bove Lab — https://bovelab.ucsf.edu
- See also: UCSF Health — https://multiplesclerosis.ucsf.edu/research

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT04002934/Prot_SAP_000.pdf